CLINICAL TRIAL: NCT00408525
Title: Efficacy of Donepezil in Normalizing Brain Activation Patterns in People Genetically at Risk for Alzheimer's Disease
Brief Title: Donepezil and Brain Activity Patterns in Those at Risk For Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 040686
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Disease
Keywords: memory loss; memory problems; alzheimer's; forgetfulness; forgetting
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Donepezil
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: donepezil — donepezil 5 mg tablets, total dose per day 10 mg for 6 week duration of study. Taken once per day.
  Other Names: Aricept

SUMMARY:
The purpose of the study is to examine patterns of brain activity in people who are at risk for memory problems (e.g., Alzheimer's disease or dementia)before and after the medication donepezil. Although genetic testing will be done, the results will not be shared with study participants.

Once the genetic testing is completed subjects may continue to the second phase of the study. During this time they will be asked to take the medication donepezil (which is approved by the FDA for the treatment of Alzheimer's disease).

Donepezil is not FDA approved for healthy volunteers and is therefore considered investigational in this study.

DETAILED DESCRIPTION:
HYPOTHESIS

1. Cognitively intact individuals with normal brain morphology at genetic risk for developing Alzheimer's' Disease (AD) show alterations in brain activation patterns during tasks that require memory compared to similar individuals with lower risk for developing AD.
2. Donepezil, a cholinesterase inhibitor, can normalize such brain activation patterns in subjects at risk for AD.

SPECIFIC AIMS

1. To replicate a recent study1, and compare brain activation in subjects genetically at risk for AD (carriers of the є4 allele of the apolipoprotein E gene (APOE)) with subjects at lower risk for AD (lacking the є4 allele) during tasks that require memory, via functional magnetic resonance imaging (fMRI).
2. To determine if administration of a drug currently indicated in the treatment of AD, donepezil, can reverse fMRI brain activation patterns of at risk subjects to patterns similar to those of subjects at lower genetic risk for AD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may report experiencing subjective memory dysfunction, however they must be found by clinical evaluation to have no memory dysfunction
* Neuropsychological test battery in the normal range
* Ages 40-85

Exclusion Criteria:

* Dementia (Mini-Mental State Exam less than 25/30)
* Left-handedness
* Current medication that could influence cognition
* Medical, psychiatric, and neurologic conditions, including cerebrovascular disease or uncontrolled hypertension
* Claustrophobia
* Surgical clips or implants
* Pacemakers or other implanted electronic devices
* History of sheet metal work

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2012-08-24 (Actual); Study Completion 2012-08-24 (Actual)

PRIMARY OUTCOMES:
Changes in brain activation patterns as measured in an fMRI. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harry E Gwirtsman, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bookheimer SY, Strojwas MH, Cohen MS, Saunders AM, Pericak-Vance MA, Mazziotta JC, Small GW. Patterns of brain activation in people at risk for Alzheimer's disease. N Engl J Med. 2000 Aug 17;343(7):450-6. doi: 10.1056/NEJM200008173430701. PMID 10944562
- [Background] Morris JC. Is Alzheimer's disease inevitable with age?: Lessons from clinicopathologic studies of healthy aging and very mild alzheimer's disease. J Clin Invest. 1999 Nov;104(9):1171-3. doi: 10.1172/JCI8560. No abstract available. PMID 10545515
- [Background] Small GW, Mazziotta JC, Collins MT, Baxter LR, Phelps ME, Mandelkern MA, Kaplan A, La Rue A, Adamson CF, Chang L, et al. Apolipoprotein E type 4 allele and cerebral glucose metabolism in relatives at risk for familial Alzheimer disease. JAMA. 1995 Mar 22-29;273(12):942-7. PMID 7884953
- [Background] Reiman EM, Caselli RJ, Yun LS, Chen K, Bandy D, Minoshima S, Thibodeau SN, Osborne D. Preclinical evidence of Alzheimer's disease in persons homozygous for the epsilon 4 allele for apolipoprotein E. N Engl J Med. 1996 Mar 21;334(12):752-8. doi: 10.1056/NEJM199603213341202. PMID 8592548
- [Background] Small GW, Ercoli LM, Silverman DH, Huang SC, Komo S, Bookheimer SY, Lavretsky H, Miller K, Siddarth P, Rasgon NL, Mazziotta JC, Saxena S, Wu HM, Mega MS, Cummings JL, Saunders AM, Pericak-Vance MA, Roses AD, Barrio JR, Phelps ME. Cerebral metabolic and cognitive decline in persons at genetic risk for Alzheimer's disease. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6037-42. doi: 10.1073/pnas.090106797. PMID 10811879
- [Background] Burggren AC, Small GW, Sabb FW, Bookheimer SY. Specificity of brain activation patterns in people at genetic risk for Alzheimer disease. Am J Geriatr Psychiatry. 2002 Jan-Feb;10(1):44-51. PMID 11790634
- [Background] Smith CD, Andersen AH, Kryscio RJ, Schmitt FA, Kindy MS, Blonder LX, Avison MJ. Women at risk for AD show increased parietal activation during a fluency task. Neurology. 2002 Apr 23;58(8):1197-202. doi: 10.1212/wnl.58.8.1197. PMID 11971086
- [Background] Padovani A, Pastorino L, Borroni B, Colciaghi F, Rozzini L, Monastero R, Perez J, Pettenati C, Mussi M, Parrinello G, Cottini E, Lenzi GL, Trabucchi M, Cattabeni F, Di Luca M. Amyloid precursor protein in platelets: a peripheral marker for the diagnosis of sporadic AD. Neurology. 2001 Dec 26;57(12):2243-8. doi: 10.1212/wnl.57.12.2243. PMID 11756604
- [Background] Borroni B, Colciaghi F, Pastorino L, Pettenati C, Cottini E, Rozzini L, Monastero R, Lenzi GL, Cattabeni F, Di Luca M, Padovani A. Amyloid precursor protein in platelets of patients with Alzheimer disease: effect of acetylcholinesterase inhibitor treatment. Arch Neurol. 2001 Mar;58(3):442-6. doi: 10.1001/archneur.58.3.442. PMID 11255448